CLINICAL TRIAL: NCT07152483
Title: The Resistant Starch Intervention for Cognitive Enhancement (RICE) in Individuals With High Genetic Risk
Brief Title: The Resistant Starch Intervention for Cognitive Enhancement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RICE
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Impairment; Diet Interventions; Cognitive Decline; Genetic Risk Factors; Obesity &Amp; Overweight
Keywords: Cognitive Impairment; Diet Interventions; Cognitive Decline; Genetic Risk Factors; Obesity & Overweight
MeSH Terms: conditions — Cognitive Dysfunction; Obesity; Overweight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-resistant starch foods intervention group (Active Comparator): Participants in the intervention group will intake high resistant starch staple foods (achieving daily intake of ≥28g resistant starch)
  Interventions: Dietary Supplement: High resistant starch staple foods
- Regular starch staple foods control group (Placebo Comparator): Participants in the control group will intake isocaloric regular starch staple foods
  Interventions: Dietary Supplement: Regular starch staple foods

INTERVENTIONS:
Dietary Supplement: High resistant starch staple foods — Participants in the intervention group will intake high resistant starch staple foods (achieving daily intake of ≥28g resistant starch)
  Arms: High-resistant starch foods intervention group
Dietary Supplement: Regular starch staple foods — Participants in the control group will intake isocaloric regular starch staple foods
  Arms: Regular starch staple foods control group

SUMMARY:
The investigation will explore the potential effects of resistant starch The Resistant Starch Intervention for Cognitive Enhancement study aimed to evaluate the effect of high-resistant starch diet intervention in slowing cognitive decline among individuals at high genetic risk for cognitive impairment. Participants will be randomly assigned to either an intervention group receiving daily high-resistant starch food products or a control group receiving isoenergetic regular starch products. The investigation will validate the potential effects of resistant starch on cognitive function protection and explore the underlying mechanisms through comprehensive data collection, including standardized neuropsychological assessments, laboratory biomarkers derived from blood and fecal specimens, and multimodal magnetic resonance imaging.

DETAILED DESCRIPTION:
The Resistant Starch Intervention for Cognitive Enhancement (RICE) in Individuals With High Genetic Risk trial is designed to evaluate the effect of high-resistant starch diet intervention in slowing cognitive decline among individuals at high genetic risk for cognitive impairment. A total of 70 participants aged ≥40 years with a meta-polygenic risk score (metaPRS) >0.4-indicating elevated genetic susceptibility-and who are overweight or abdominally obese, will be randomly assigned in a 1:1 ratio to either an intervention group receiving daily high-resistant starch food products (≥28 g/day) or a control group receiving isoenergetic regular starch products. The investigation will validate the potential effects of resistant starch on cognitive function protection and explore the underlying mechanisms through comprehensive data collection, including standardized neuropsychological assessments, laboratory biomarkers derived from blood and fecal specimens, and multimodal magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 40 years
* meta-polygenic risk score (metaPRS) > 0.4
* Montreal Cognitive Assessment (MoCA) score ≤ 26
* Central obesity (waist circumference > 90 cm in males or > 80 cm in females) or body mass index (BMI) ≥ 28 kg/m²
* Written informed consent available
* Proficient in using smartphones
* Willingness to complete all assessments and participate in follow-up

Exclusion Criteria:

* Known hypersensitivity or allergy to resistant starch
* previously diagnosed dementia
* Suspected dementia after clinical assessment by study physician at screening visit
* Previous history of major head trauma and any intracranial surgery
* Intracranial abnormalities, such as intracerebral hemorrhage, subarachnoid hemorrhage and other space occupying lesions
* Extrapyramidal symptoms or mental illness which may affect neuropsychological measurement
* Severe loss of vision, hearing, or communicative ability
* Patients presenting a malignant disease with life expectancy < 3 years
* Participation in an ongoing investigational drug study
* The participant or a first-degree relative is currently participating in another clinical trial involving nutritional intervention.

Exit Criteria:

* Not meet the inclusion criteria
* For any poor adherence, not comply with the requirements of the follow-up, or safety reasons determined by investigator
* Any adverse or serious adverse events during the study period judged by Investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 6 months
  Primary Outcome

SECONDARY OUTCOMES:
Cognitive domain change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 6 months
  Secondary Outcome
Cognitive function change assessed by Montreal Cognitive Assessment (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 6 months
  Secondary Outcome
Gut microbiota determined by measuring specific bacterial levels in the fecal samples | 6 months
  Secondary Outcome
Metabolite composition to measure the metabolite profiles in participants' faecal samples and serum samples | 6 months
  Secondary Outcome
Change in waist circumference | 6 months
  Secondary Outcome
Change in body mass index (BMI) | 6 months
  Secondary Outcome
Changes in glymphatic function assessed by dispersion coefficient of periarterial and perivenous spaces on diffusion tensor imaging (DTI) | 6 months
  Secondary Outcome
Changes in image markers (white matter hyperintensity, lacunes, microbleeds, perivascular spaces, brain atrophy, micro-infarcts) of CSVD assessed on MRI | 6 months
  Secondary Outcome
Changes in brain functional network connectivity assessed by resting state functional magnetic resonance imaging (fMRI) | 6 months
  Secondary Outcome
Global cognitive function change assessed with Z-score of a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months
  Secondary Outcome
Working memory domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months
  Secondary Outcome
Executive function domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months
  Secondary Outcome
Language domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months
  Secondary Outcome
Visual motor speed domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months
  Secondary Outcome
Visual spatial function domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months
  Secondary Outcome
Memory and recognition domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months
  Secondary Outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affilated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No